CLINICAL TRIAL: NCT00004645
Title: Phase III Randomized, Double-Blind, Sham-Controlled Study of Plasma Exchange for Acute Severe Attacks of Inflammatory Demyelinating Disease Refractory to Intravenous Methylprednisolone
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: Mayo Clinic (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/11693; MAYOC-29493
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-03

CONDITIONS: Acute Disseminated Encephalomyelitis; Devic's Syndrome; Marburg's Variant of Multiple Sclerosis; Balo's Concentric Sclerosis; Acute Transverse Myelitis
Keywords: Balo's concentric sclerosis; Devic's syndrome; Marburg's variant of multiple sclerosis; acute disseminated encephalomyelitis; acute transverse myelitis; multiple sclerosis; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Encephalomyelitis, Acute Disseminated; Neuromyelitis Optica; Diffuse Cerebral Sclerosis of Schilder; Myelitis, Transverse; Multiple Sclerosis; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Plasma Exchange

INTERVENTIONS:
Procedure: Plasma exchange

SUMMARY:
OBJECTIVES:

I. Evaluate the effectiveness of plasma exchange in the treatment of acute severe attacks of inflammatory demyelinating disease in patients who have failed intravenous steroid therapy.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double-blind study. Patients are stratified by disease type; each stratum is randomized separately.

The first group of patients receives a true plasma exchange using continuous-flow centrifugation with serum albumin and crystalloid replacement every 2 days for a total of 7 exchanges.

The second group receives a sham plasma exchange with no centrifugation every 2 days for a total of 7 exchanges.

Patients cross to the alternate therapy if there is less than a moderate improvement by day 14. The treatment decision is based on a blinded neurologic assessment.

Concurrent corticosteroids and other immunosuppressants, and high-dose barbiturates are not allowed.

Patients are followed at 1 and 6 months after the last exchange.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Idiopathic inflammatory demyelinating syndrome, as follows: biopsy-proven if necessary - established diagnosis of multiple sclerosis (MS) using Poser criteria; acute disseminated encephalomyelitis; Marburg's variant of MS Balo's concentric sclerosis
* Eligible without biopsy: acute transverse myelitis; Devic's syndrome
* Acute neurologic deficit markedly affecting consciousness, language, or brainstem/spinal cord function, i.e., aphasia, paraplegia, coma, quadriplegia, hemiplegia, severe organic brain syndrome
* Deficit unresponsive to 5 days of high-dose intravenous methylprednisolone (MePRDL), as follows: deficit duration of 21 days to 3 months AND no improvement 14 days after beginning MePRDL OR deficit duration of 12 to 20 days AND continued deterioration after completion of MePRDL
* No chronically progressive demyelinating disease
* No HIV-associated demyelinating syndrome
* No progressive multifocal leukoencephalopathy
* No optic neuritis

--Prior/Concurrent Therapy--

* No more than 3 months of prior steroid therapy Failure on prior MePRDL required Minimum dose 7 mg/kg per day for 5 days
* At least 6 weeks since other immunosuppressives, e.g., cyclophosphamide, azathioprine, cyclosporine

--Patient Characteristics--

* Renal: Creatinine less than 1.5 mg/dL
* Cardiovascular: No hypovolemia; no infarction; no vasculitis; no other major systemic cardiovascular illness
* Pulmonary: No major respiratory illness
* Other: No infection, including hepatitis or human immunodeficiency virus; no recent intravenous drug abuse; no high-risk sexual behavior; no cardiac, cerebrovascular, or autonomic dysfunction that would increase risk of hypotension; no other major systemic illness that would preclude protocol therapy; no pregnant or nursing women; negative serum pregnancy test required of fertile women; effective contraception required

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22
Dates: Start 1995-01

CONTACTS AND LOCATIONS:
Overall Officials: Brian G. Weinshenker, Study Chair — Mayo Clinic